CLINICAL TRIAL: NCT06002516
Title: The RELIEF-pathway in Patients With Upper Abdominal Pain; an Open-label Multicenter Randomized Controlled Trial
Brief Title: RELIEF-pathway in Patients With Upper Abdominal Pain
Acronym: RELIEF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-12618
Record Dates: First submitted 2023-08-07; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Abdominal Pain; Gallstone; Colic; Dyspepsia; Irritable Bowel Syndrome; Health Care Utilization; Patient Reported Outcomes; Upper Abdominal Pain; Decision Aid
Keywords: Abdominal pain; Health care utilization
MeSH Terms: conditions — Abdominal Pain; Gallstones; Colic; Dyspepsia; Irritable Bowel Syndrome; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled open-label superiority trial, with two parallel arms, usual care (control arm) versus the RELIEF pathway (intervention arm). Patients will randomly be assigned (1:1) to usual care or the RELIEF pathway with use of stratification for disease severity, age and sex.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RELIEF pathway (Experimental): Patients in the intervention group (RELIEF-pathway) will receive access to the web-based education tool before visit of the outpatient clinic of Surgery or Gastroenterology.
  Interventions: Other: RELIEF-pathway
- Usual care (No Intervention): Patients assigned to the control group will receive the usual care given at participating centers. During the first visit at the surgery or gastroenterology outpatient clinic subjects are seen by a random medical specialist, who will assess history, examine the patient, and review investigations. Diagnostic and treatment decisions will be based on the physician's preference and experience and on the patients' preferred choice of treatment.

INTERVENTIONS:
Other: RELIEF-pathway — The personalized web-based education tool contains information on:
  * Information of cause and symptoms of functional dyspepsia, irritable bowel syndrome and uncomplicated symptomatic cholecystolithiasis;
  * Symptom checker based on the ROME III and ROME IV criteria;
  * Red flags symptoms defined as direct or indirect signs of upper GI hemorrhage.
  * Lifestyle adjustments to improve abdominal symptoms and quality of life.
  * Information on effect of upper gastrointestinal endoscopy, colonoscopy and laparoscopic cholecystectomy.
  After the web-based education tool is completed we will offer an additional visit at the Prevention and Lifestyle clinic, this is optional and not obligatory.
  Arms: RELIEF pathway

SUMMARY:
Upper abdominal pain (UAP) is a common symptom and frequently the reason to visit the hospital. The prevalence of epigastric pain in the Dutch population is estimated to be as high as 37%. Moreover, Dutch hospitals yearly record >100.000 diagnoses related to UAP. In most patients, UAP can be attributed to symptomatic (functional) dyspepsia (FD), Irritable Bowel Syndrome (IBS) or uncomplicated gallstone disease (cholecystolithiasis), with a prevalence in the general population of 20-30%, 20%, and 6-9%, respectively. However, these conditions may have overlapping symptom patterns and generally affect similar populations. which contributes to ineffective (diagnostic) interventions. Patients are generally not aware of the similarity of symptoms and the poor outcome of some treatments.

Education positively influences patients' self-management and health judgment. In a recent open-label, multicentre trial the effectiveness of web-based patients' education is applied to reduce overuse of upper gastrointestinal endoscopies in patients with dyspepsia. This study illustrated that an web-based education tool safely reduced 40% in upper gastrointestinal endoscopies. Lifestyle interventions (such as change of diet and/or physical activity) are widely incorporated in treatment programs for cardio-vascular diseases including diabetes mellitus and obesity. An web-based education tool on upper abdominal pain and other complaints combined with a lifestyle interventions for patients may be an effective treatment option for this large group of patients.

This study investigates the potential of an individualized web-based education tool as intervention for patients with functional dyspepsia, irritable bowel syndrome and uncomplicated symptomatic cholecystolithiasis with the possibility to visit the Prevention and Lifestyle clinic (RELIEF pathway). The RELIEF pathway aims to reduce unnecessary health care utilization and, secondly, to maintain and improve quality of life by educating patients on lifestyle improvement.

DETAILED DESCRIPTION:
Objective: The main goal is to evaluate the effect of the RELIEF pathway versus usual care on health care utilization in terms of hospital visits and number of interventions.

Study design: A multicenter randomized controlled open-label superiority trial, with two parallel arms, usual care (control arm) versus the RELIEF pathway (intervention arm). Patients will randomly be assigned (1:1) to usual care or the RELIEF pathway with use of stratification for disease severity, age and sex.

Study population: All patients between 18 and 70 years old, with a first referral by their general practitioner (GP) to the Department of Surgery or Gastroenterology with functional dyspepsia (ICPC D87.02), irritable bowel syndrome (ICPC D93) or uncomplicated symptomatic cholecystolithiasis (ICPC D98.03). Patients are not eligible for inclusion if they and/or GP report alarm symptoms, which may be direct or indirect signs of cancer or upper GI tract bleeding: weight loss, persistent vomiting, dysphagia, jaundice, hematemesis, melena, haematochezia, or anaemia. Patients with a first or second-degree relative with a history of upper GI tract malignant neoplasm, patients with a history of complicated cholecystolithiasis (acute cholecystitis, choledocholithiasis, biliary pancreatitis and cholangitis) or a history of or current malignancy (except SCC or BCC of the skin).

Intervention:

Patients in the intervention group (RELIEF-pathway) will receive access to the web-based education tool before visit of the outpatient clinic of Surgery or Gastroenterology.

The personalized web-based education tool contains information on:

* Information of cause and symptoms of functional dyspepsia, irritable bowel syndrome and uncomplicated symptomatic cholecystolithiasis;
* Symptom checker based on the ROME III and ROME IV criteria;
* Red flags symptoms defined as direct or indirect signs of upper GI hemorrhage.
* Lifestyle adjustments to improve abdominal symptoms and quality of life.
* Information on effect of upper gastrointestinal endoscopy, colonoscopy and laparoscopic cholecystectomy.

The investigators aim that the patient will complete the web-based education tool before visiting the outpatient clinic of Surgery and Gastroenterology. The web-based education tool is available during 12 months after randomization.

After the web-based education tool is completed we will offer an additional visit at the Prevention and Lifestyle clinic, this is optional and not obligatory.

Control: Patients assigned to the control group will receive the usual care given at participating centers. During the first visit at the surgery or gastroenterology outpatient clinic subjects are seen by a random medical specialist, who will assess history, examine the patient, and review investigations.Diagnostic and treatment decisions will be based on the physician's preference and experience and on the patients' preferred choice of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years old.
* First referral due to upper abdominal pain (UAP) and symptoms due to Functional dyspepsia (ICPC code 87.02), Irritable Bowel syndrome (ICPC 93.0) or uncomplicated symptomatic cholecystolithiasis (ICPC 98.03).
* Proficient in reading and understanding of the Dutch language.
* Referred to the outpatient clinic of gastroenterology or surgery.
* Providing informed consent.

Exclusion Criteria:

* If the following alarm symptoms are reported in the referral letter by the GP: weight loss, persistent vomiting, dysphagia, jaundice, hematemesis, melena, haematochezia, or anaemia.
* Any other direct or indirect signs of cancer or upper GI tract bleeding.
* Patients with a first or second-degree relative with a history of upper GI tract malignant neoplasm.
* Patients with a history of complicated cholecystolithiasis.
* A history of or current malignancy (except SCC or BCC of the skin).
* Pregnancy;
* Expected short life span of less than 12 months.
* Known cirrhosis of the liver
* Current schizophrenia, memory deficiency, or any other disorder that predispose them to unreliable questionnaire responses;
* Mentally incompetent;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | 6 months
  Healthcare-utilization regarding to upper abdominal pain:
  * Number of outpatient clinics regarding to UAP
  * Number of diagnostics (Upper GI endoscopies, colonoscopies).
  * Number of treatments (laparoscopic cholecystectomy).
  * Number of ER visits.
  Medical records will be evaluated on above mentioned points.

SECONDARY OUTCOMES:
Patient-reported outcomes | 12 months
  Assessed by the following questionnaires:
  * ROME III criteria for biliary colic (ROMEIII)
  * ROME IV criteria for FGID (ROMEIV))
  * Hospital anxiety and depression scale (HADS questionnaire)
  * Symptom severity (PAGI-SYM questionnaire).
  * Short-Form Health and Labour Questionnaire (SF-HLQ questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis van Laarhoven, MD PhD, Principal Investigator — Radboud University Medical Center

REFERENCES:
- [Background] de Jong JJ, Lantinga MA, Tan ACITL, Aquarius M, Scheffer RCH, Uil JJ, de Reuver PR, Keszthelyi D, Westert GP, Masclee AAM, Drenth JPH. Web-Based Educational Intervention for Patients With Uninvestigated Dyspepsia Referred for Upper Gastrointestinal Tract Endoscopy: A Randomized Clinical Trial. JAMA Intern Med. 2021 Jun 1;181(6):825-833. doi: 10.1001/jamainternmed.2021.1408. PMID 33900373
- [Background] van Dijk AH, Wennmacker SZ, de Reuver PR, Latenstein CSS, Buyne O, Donkervoort SC, Eijsbouts QAJ, Heisterkamp J, Hof KI', Janssen J, Nieuwenhuijs VB, Schaap HM, Steenvoorde P, Stockmann HBAC, Boerma D, Westert GP, Drenth JPH, Dijkgraaf MGW, Boermeester MA, van Laarhoven CJHM. Restrictive strategy versus usual care for cholecystectomy in patients with gallstones and abdominal pain (SECURE): a multicentre, randomised, parallel-arm, non-inferiority trial. Lancet. 2019 Jun 8;393(10188):2322-2330. doi: 10.1016/S0140-6736(19)30941-9. Epub 2019 Apr 27. PMID 31036336
- [Background] Kok L, Elias SG, Witteman BJ, Goedhard JG, Romberg-Camps MJ, Muris JW, Moons KG, de Wit NJ. Application of the Rome III criteria is not likely to reduce the number of unnecessary referrals for colonoscopy in primary care. Eur J Gastroenterol Hepatol. 2013 May;25(5):568-74. doi: 10.1097/MEG.0b013e32835d4ddd. PMID 23325277
- [Background] Latenstein CSS, Hannink G, van der Bilt JDW, Donkervoort SC, Eijsbouts QAJ, Heisterkamp J, Nieuwenhuijs VB, Schreinemakers JMJ, Wiering B, Boermeester MA, Drenth JPH, van Laarhoven CJHM, Dijkgraaf MGW, de Reuver PR; SECURE trial collaborators. A Clinical Decision Tool for Selection of Patients With Symptomatic Cholelithiasis for Cholecystectomy Based on Reduction of Pain and a Pain-Free State Following Surgery. JAMA Surg. 2021 Oct 1;156(10):e213706. doi: 10.1001/jamasurg.2021.3706. Epub 2021 Oct 13. PMID 34379080
- [Background] de Jong JJ, Latenstein CSS, Boerma D, Hazebroek EJ, Hirsch D, Heikens JT, Konsten J, Polat F, Lantinga MA, van Laarhoven CJHM, Drenth JPH, de Reuver PR. Functional Dyspepsia and Irritable Bowel Syndrome are Highly Prevalent in Patients With Gallstones and Are Negatively Associated With Outcomes After Cholecystectomy: A Prospective, Multicenter, Observational Study (PERFECT - Trial). Ann Surg. 2022 Jun 1;275(6):e766-e772. doi: 10.1097/SLA.0000000000004453. Epub 2020 Sep 1. PMID 32889877